CLINICAL TRIAL: NCT07169630
Title: PET Imaging of Phosphodiesterase-4 (PDE4) in Volunteers With Alzheimer s Disease (AD) or Mild Cognitive Impairment (MCI)
Brief Title: PET Imaging of Phosphodiesterase-4 (PDE4) in Volunteers With Alzheimer Disease (AD) or Mild Cognitive Impairment (MCI)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10002277; 002277-M
Record Dates: First submitted 2025-09-11; First posted 2025-09-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-05

CONDITIONS: Alzheimer s Disease; Mild Cognitive Impairment; Healthy
Keywords: 18F-PF-06445974; PET Imaging
MeSH Terms: conditions — Cognitive Dysfunction | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- One-Arm (Other): All subjects will receive the same tests.
  Interventions: Drug: 18F-PF974; Drug: 18F-florbetaben

INTERVENTIONS:
Drug: 18F-PF974 — Injected IV followed by PET scanning
Drug: 18F-florbetaben — Injected IV followed by PET scanning

SUMMARY:
Background:

About 5 million adults in the United States have age-related brain disorders. These include Alzheimer disease (AD), mild cognitive impairment (MCI), and other dementias. The number of people with these disorders will likely increase as the population ages and life span increases. Inflammation is thought to play a role in AD and MCI. Researchers want to know if an enzyme called PDE4B increases inflammation in people with AD or MCI.

Objective:

To test whether medical imaging using a new radiotracer ([18F]PF-06445974) can measure PDE4B in the brains of people with AD or MCI.

Eligibility:

People aged 50 years and older with AD or MCI. Healthy volunteers are also needed.

Design:

Participants will have up to 5 clinic visits with 3 imaging scans of the brain.

They will have be screened. They will have a physical exam with blood tests. This will include tests of their heart and nerve function, including memory.

Participants will have 2 positron emission tomography (PET) scans. One will use a standard radiotracer. The other will use the study radiotracer. They will receive each tracer through a tube attached to a needle inserted into a vein. During the scan with the study tracer, participants will have a second tube inserted into a vein in the wrist; this tube will be used to draw blood during the scan. Participants will lie on a bed that slides into a doughnut-shaped machine. These visits will take about 6 hours each.

Participants will have 1 magnetic resonance imaging (MRI) scan. They will lie on a bed that slides into a cylinder. This visit will take up to 2 hours....

DETAILED DESCRIPTION:
Study Description:

As a biomarker of neuroinflammation, the density of PDE4B is hypothesized to be elevated in individuals with AD or MCI compared to age-matched healthy volunteers (HVs). Participants will receive two positron emission tomography (PET) scans (for PDE4B and for beta-amyloid (A beta)) and one magnetic resonance imaging (MRI) scan of the brain.

Objectives:

Primary Objective:

To determine whether PDE4B radioligand binding is increased in medial temporal lobe of participants with AD or MCI (both A beta positive) compared to age-and sex matched HVs (who are A beta negative)

Exploratory Objective #1:

To determine whether PDE4B binding in the medial temporal lobe is correlated with demographic variables, clinical markers, or biological markers.

Exploratory Objective #2:

To determine whether any region of the brain in individuals with AD or MCI has increased PDE4B binding compared to HVs.

Endpoints:

Primary endpoints: PET measurements of PDE4B; clinical variables, including neuropsychological tests; and biological variables, including plasma concentrations of A(beta)40, A(beta)42, total tau, and Ptau217.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be referred by a physician with the suspected diagnosis of AD or MCI. However, the PI of this protocol will provide the final diagnosis. For this reason, this protocol will have just one consent form for participants suspected of having either AD or MCI.

AD and MCI Study Groups:

Participants must meet all the following criteria:

* Aged 50 or older.
* Be able (or have their Legally Authorized Representative (LAR) be able) to understand the study and be willing to sign a written informed consent document.
* Have been diagnosed by a neurologist or psychiatrist with MCI or AD.
* Be in good general health as evidenced by medical history and physical examination.
* Have had their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
* Agree to adhere to the lifestyle considerations.

Healthy Volunteers:

Participants must meet all the following criteria:

* Aged 50 or older.
* Able to provide informed consent.
* Be in good general health, as evidenced by medical history and physical examination, and have no cognitive impairment.
* Have had their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
* Agree to adhere to the lifestyle considerations.

EXCLUSION CRITERIA:

Both the study groups will be excluded if they meet any of the following criteria:

* Clinically significant abnormalities on EKG or laboratory testing. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen).
* Participants should not have taken non-steroidal anti-inflammatory drugs (NSAIDs) for two weeks prior to the PET scan. Aspirin, corticosteroids (with the exception of skin products), or immunosuppressants (e.g., methotrexate) must not have been taken in the prior month.
* Have other major neurological or medical diseases that may cause cognitive dysfunction, such as structural brain diseases, metabolic diseases, paraneoplastic syndromes, infectious diseases, or other significant neurological abnormalities.
* Have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
* Are unable to travel to the NIH.
* Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
* Have an inability to lie flat and/or lie still on the camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the volunteer and/or caregiver during the screening visit.
* Participants must not have substance use disorder or alcohol use disorder.
* Participants should not be under treatment or previously treated with an amyloid antibody such as lecanemab.
* Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye).
* Pregnancy or breast feeding.
* HIV infection.
* Non-English speaking participants.

Exclusion of Children:

Inclusion of children is not appropriate, because this protocol has more than minimal risk from radiation exposure without the possibility of direct benefit.

Exclusion of Pregnant or Breastfeeding Women:

Pregnant women will be excluded because this protocol involves exposure to ionizing radiation. Lactating women will be excluded because radioisotopes may be excreted in milk. We will not require contraception for this protocol to allow participants autonomy in medical decision-making. However, while we will not require contraception for woman of childbearing potential, we will perform a pregnancy test at screening and prior to all procedures to ensure participants are not pregnant

Exclusion of Participants who are HIV Positive:

Persons with HIV infection are excluded because HIV infection itself may change cAMP signaling.

Exclusion of Non-English-Speaking Participants:

Non-English-speaking participants will be excluded from participation in this study because neuropsychological testing is required by this protocol. This testing, which is critical for interpreting study results, has not been validated in other languages or when using a translator.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2029-04-11 (Estimated); Study Completion 2030-04-11 (Estimated)

PRIMARY OUTCOMES:
To determine whether PDE4B radioligand binding is increased in medial temporal lobe of participants with AD or MCI (both A <= positive) compared to age-and sex matched HVs (who are A <= negative. | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Parcon, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The results will be submitted to ClinicalTrials.gov
Supporting Information: Study Protocol
Time Frame: 18 months after closure of protocol.
Access Criteria: BTRIS

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002277-M.html